CLINICAL TRIAL: NCT00988221
Title: A 24 Week Randomized, Double-blind, Placebo-controlled Withdrawal Trial With a 16 Week Open-label lead-in Phase, and 64 Week Open-label Follow-up, to Evaluate the Effect on Clinical Response and the Safety of Tocilizumab in Patients With Active Polyarticular-course Juvenile Idiopathic Arthritis
Brief Title: A Study of Tocilizumab in Patients With Active Polyarticular Juvenile Idiopathic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA19977; 2009-011593-15 (EudraCT Number)
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2012-11-01 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-06

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Tocilizumab 10 mg/kg in patients weighing < 30 kg (Experimental): Patients received tocilizumab 10 mg/kg intravenously every 4 weeks.
  Interventions: Drug: Tocilizumab
- Tocilizumab 8 mg/kg in patients weighing < 30 kg (Experimental): Patients received tocilizumab 8 mg/kg intravenously every 4 weeks.
  Interventions: Drug: Tocilizumab
- Tocilizumab 8 mg/kg in patients weighing ≥ 30 kg (Experimental): Patients received tocilizumab 8 mg/kg intravenously every 4 weeks.
  Interventions: Drug: Tocilizumab
- Placebo (Placebo Comparator): Patients received placebo to tocilizumab intravenously every 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab was supplied as a sterile solution in vials.
  Other Names: RoActemra; Actemra
  Arms: Tocilizumab 10 mg/kg in patients weighing < 30 kg; Tocilizumab 8 mg/kg in patients weighing < 30 kg; Tocilizumab 8 mg/kg in patients weighing ≥ 30 kg
Drug: Placebo — Placebo to tocilizumab was supplied as a sterile solution in vials.
  Arms: Placebo

SUMMARY:
This 3-part study evaluated the efficacy and safety of tocilizumab in patients with active polyarticular-course juvenile idiopathic arthritis who have an inadequate response to, or were intolerant of methotrexate. In Part I of the study, all patients received intravenous (iv) infusions of tocilizumab (8 mg/kg for patients ≥ 30kg, 8 mg/kg or 10 mg/kg for patients < 30kg) every 4 weeks for 16 weeks. In Part II of the study, patients with an adequate response in Part I were randomized to receive either tocilizumab at the same dose as in Part I or placebo every 4 weeks for up to 24 weeks. In Part III of the study, patients received tocilizumab at the same dose as in Part I every 4 weeks for up to another 64 weeks. Standard of care therapy with or without non-steroidal anti-inflammatory drugs (NSAID), corticosteroids, or methotrexate was continued throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Children/juveniles, 2-17 years of age.
* Polyarticular-course juvenile idiopathic arthritis (pcJIA) ≥ 6 months duration.
* Active disease (≥ 5 active joints, ≥ 3 with limitation of motion).
* Inadequate response to or inability to tolerate methotrexate.
* Methotrexate, oral corticosteroids, and non-steroidal anti-inflammatory drugs (NSAID) at stable dose(at least 8, 4, and 2 weeks,respectively) prior to baseline.
* Biologics discontinued, between at least 1 and 20 weeks prior to baseline, depending on biologic.

Exclusion Criteria:

* Auto-immune, rheumatic disease or overlap syndrome other than pcJIA.
* Wheelchair bound or bedridden.
* Intra-articular, intramuscular, intravenous, or long-acting corticosteroids within 4 weeks prior to baseline.
* Disease-modifying anti-rheumatic drugs (DMARD) (other than methotrexate) within 4 weeks prior to baseline.
* Previous treatment with tocilizumab.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2009-11-30 (Actual); Primary Completion 2011-11-30 (Actual); Study Completion 2013-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (69):
- United States (10):
  - Connecticut Children's Medical Center; 5E Clinical Trials Unit, Hartford, Connecticut
  - Children's National Medical Center; Pediatric Rheumatology, Washington D.C., District of Columbia
  - Delray Research Associates, Delray Beach, Florida
  - Miami Children's Hospital, Miami, Florida
  - The University of Chicago;Department of Pediatrics, Chicago, Illinois
  - University of Louisville Research Foundation, Inc; Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Children's Hospital, New Orleans, Louisiana
  - Hackensack University Medical Center; Pediatric Rheumatology, Hackensack, New Jersey
  - Cincinnati Children'S Hospital Medical Center; Division of Rheumatology, Cincinnati, Ohio
  - Healthcare Research Consultants, Tulsa, Oklahoma
- Argentina (4):
  - Hospital Gral de Niños Pedro Elizalde, Buenos Aires
  - Hospital de Niños; Reumatologia, Buenos Aires
  - Caici; Rheumatology, Rosario
  - Centro Medico Privado de Reumatologia; Reumathology, San Miguel
- Australia (3):
  - Westmead Hospital; Paediatric Rheumatology, Westmead, New South Wales
  - Royal Children'S Hospital; Paediatric Rheumatology, Parkville, Victoria
  - Princess Margaret Children'S Hospital; Department of Immunology, Subiaco, Western Australia
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Brazil (4):
  - Hospital Universitario Pedro Ernesto; Nucleo de Estudos da Saude do Adolescente, Rio de Janeiro, Rio de Janeiro
  - Instituto de Puericultura E Pediatria Martagão Gesteira, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - FMUSP; Instituto da Crianca - Reumatologia, São Paulo, São Paulo
- Canada (4):
  - Alberta Children'S Hospital, Calgary, Alberta
  - British Columbia Children's Hospital; Rheumatology, Vancouver, British Columbia
  - Children'S Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital For Sick Children, Toronto, Ontario
- France (6):
  - Hôpital Pellegrin; Urgences Pédiatriques, Bordeaux
  - CH de Bicêtre; Pediatrie Generale, Le Kremlin-Bicêtre
  - Hôpital Lapeyronie; Immuno-Rhumatologie Pr Jorgensen, Montpellier
  - Hopital Cochin; Rhumatologie A, Paris
  - Hop Necker Enfants Malades;UIH, Paris
  - Hopitaux De Brabois; Medecine Infantile II, Vandœuvre-lès-Nancy
- Germany (4):
  - Charité Campus; Virchow Klinikum Berlin, Berlin
  - Klinik Bremen-Mitte; Prof. Hess-Kinderklinik, Bremen
  - Clementine Hospital; Kinder- und Jugendrheumatologie, Frankfurt am Main
  - Asklepios Klinik; Zentrum fuer Allgemeine Paediatrie und Neonatologie, Sankt Augustin
- Italy (5):
  - Irccs Ospedale Pediatrico Bambin Gesu - Dip. Di Medicina, Rome, Lazio
  - IRCCS G. Gaslini; Pediatria II, Genoa, Liguria
  - ASST CENTRO SPECIALISTICO ORTOPEDICO TRAUMATO-LOGICO GAETANO PINI/CTO; Reumatol. Pediatrica, Milan, Lombardy
  - Nuovo Ospedale Pediatrico Meyer; Reumatologia - Clinica Pediatrica 1°, Florence, Tuscany
  - Univ. Di Padova - Dip. Di Pediatria - Unita' Reumatol. Pediatrica, Padua, Veneto
- Mexico (4):
  - Inst. Mexicano de Investigacion Clinica, Mexico City
  - Cif Biotec Medica Sur, Mexico City, Distrito Federal
  - Cliditer SA de CV, Miexico City
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez; Pediatria, Monterrey
- Peru (3):
  - Clinica San Felipe; Consultorio de Reumatología, Lima
  - Clinica San Borja; Servicio De Reumatologia, Lima
  - Instituto Nacional De Salud Del Niño, Lima
- Poland (6):
  - Wojewodzki Szpital Dzieciecy Im. J. Brudzinskiego, Bydgoszcz
  - Wojewodzki Specjalistyczny Szpital Dzieciecy Sw Ludwika; Oddzial Dzieci Starszych, Krakow
  - Uniwersytecki Szpital Kliniczny Nr 4 im. M. Konopnickiej; Oddz. Kardiolog. i Reumatolog. dla Dzieci, Lodz
  - Dzieciecy Szpital Kliniczny IM. Prof. A. Gebali; Oddzial Pediatrii Chorob Pluc I Reumatologii, Lublin
  - Centrum Pediatrii im Jana Pawla II; Oddzial Reumatologiczny, Sosnowiec
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. Prof. Eleonory Reicher, Warsaw
- Russia (6):
  - FSBI "Scientific Research Institute of Rheumatology" of russian Academy of Medical Sciences, Moscow
  - SI Sceintific children health center RAMS, Moscow
  - I. M. Sechenov Moscow State Medical University; The Ministry of Health and Social Development of RF, Moscow
  - Southern District Medical Center of Roszdrav, Rostov-on-Don
  - Saint-Petersburg State; Pediatrics Medical Academy, Saint Petersburg
  - Samara Regional Clinical Cardiology Dispensary, Samara
- Spain (5):
  - Hospital Universitario Reina Sofia; Servicio de Reumatologia, Córdoba
  - Hospital General Universitario Gregorio Marañon; Servicio de Reumatología, Madrid
  - Hospital Ramon y Cajal ; Servicio de Reumatologia, Madrid
  - Hospital Universitario Virgen Macarena; Servicio de Reumatologia, Seville
  - Hospital Universitario la Fe: Servicio de Reumatologia Pediatrica, Valencia
- United Kingdom (3):
  - Bristol Royal Hospital For Children, Bristol
  - Royal Liverpool Childrens Hospital; Rheumatology, Liverpool
  - Great Ormond Street Hospital for Sick Children; Institute of Child Health, London

REFERENCES:
- [Derived] Lim LSH, Lokku A, Pullenayegum E, Ringold S. Probability of Response in the First Sixteen Weeks After Starting Biologics: An Analysis of Juvenile Idiopathic Arthritis Biologics Trials. Arthritis Care Res (Hoboken). 2023 Jun;75(6):1238-1249. doi: 10.1002/acr.25003. Epub 2023 Jan 18. PMID 36651601
- [Derived] Malattia C, Ruperto N, Pederzoli S, Palmisani E, Pistorio A, Wouters C, Dolezalova P, Flato B, Garay S, Giancane G, Wells C, Douglass W, Brunner HI, De Benedetti F, Ravelli A; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG). Tocilizumab may slow radiographic progression in patients with systemic or polyarticular-course juvenile idiopathic arthritis: post hoc radiographic analysis from two randomized controlled trials. Arthritis Res Ther. 2020 Sep 10;22(1):211. doi: 10.1186/s13075-020-02303-y. PMID 32912276
- [Derived] Pardeo M, Wang J, Ruperto N, Alexeeva E, Chasnyk V, Schneider R, Horneff G, Huppertz HI, Minden K, Onel K, Zemel L, Martin A, Kone-Paut I, Siamopoulou-Mavridou A, Silva CA, Porter-Brown B, Bharucha KN, Brunner HI, De Benedetti F; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG). Neutropenia During Tocilizumab Treatment Is Not Associated with Infection Risk in Systemic or Polyarticular-course Juvenile Idiopathic Arthritis. J Rheumatol. 2019 Sep;46(9):1117-1126. doi: 10.3899/jrheum.180795. Epub 2019 Mar 1. PMID 30824645
- [Derived] Brunner HI, Ruperto N, Zuber Z, Keane C, Harari O, Kenwright A, Lu P, Cuttica R, Keltsev V, Xavier RM, Calvo I, Nikishina I, Rubio-Perez N, Alexeeva E, Chasnyk V, Horneff G, Opoka-Winiarska V, Quartier P, Silva CA, Silverman E, Spindler A, Baildam E, Gamir ML, Martin A, Rietschel C, Siri D, Smolewska E, Lovell D, Martini A, De Benedetti F; Paediatric Rheumatology International Trials Organisation PRINTO; Pediatric Rheumatology Collaborative Study Group (PRCSG). Efficacy and safety of tocilizumab in patients with polyarticular-course juvenile idiopathic arthritis: results from a phase 3, randomised, double-blind withdrawal trial. Ann Rheum Dis. 2015 Jun;74(6):1110-7. doi: 10.1136/annrheumdis-2014-205351. Epub 2014 May 16. PMID 24834925

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Part I, patients received either tocilizumab 8 or 10 mg/kg. In Part II, eligible patients were randomized to receive placebo or the same dose of tocilizumab as in Part I of the study. In Part III, patients received the same dose of tocilizumab as in Part I of the study, with adjustments based on weight and change in weight from Baseline.
Period: Part I
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Placebo
Started | 35 | 34 | 119 | 0 (No patients received placebo in Part I of this study.)
Completed | 31 | 24 | 111 | 0
Not Completed | 4 | 10 | 8 | 0
Not completed — Adverse Event | 0 | 1 | 2 | 0
Not completed — Insufficient Therapeutic Response | 4 | 6 | 5 | 0
Not completed — Refused Treatment | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: Part II
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Placebo
Started | 16 (Some of the patients in this group in Part I were randomized to receive placebo in Part II.) | 11 (Some of the patients in this group in Part I were randomized to receive placebo in Part II.) | 55 (Some of the patients in this group in Part I were randomized to receive placebo in Part II.) | 84
Completed | 15 | 11 | 52 (One participant who did not complete Part II was available to continue in the study and did.) | 81
Not Completed | 1 | 0 | 3 | 3
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2
Not completed — Reason not Specified | 0 | 0 | 1 | 0
Period: Part III
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Placebo
Started | 30 | 24 | 106 | 0 (No patients received placebo in Part III of this study.)
Completed | 29 | 23 | 103 | 0
Not Completed | 1 | 1 | 3 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Insufficient Therapeutic Response | 0 | 1 | 1 | 0
Not completed — Refused Treatment | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Total
Number analyzed (Participants) | 35 | 34 | 119 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.9 (3.02) | 7.6 (2.71) | 13.1 (2.78) | 11.0 (4.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 24 | 90 | 144
  Male | 5 | 10 | 29 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With a Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology 30 (ACR30) Flare in Part II of the Study (Weeks 16-40)
Description: JIA ACR30 flare is defined as a ≥ 30% worsening of 3 of 6 variables and no more than 1 of the remaining variables improving > 30%. The 6 variables are physician global assessment of disease activity (worsening of 20 units minimum on a 0-100 visual analog scale [VAS]), parent/patient global assessment of overall well-being (worsening of 20 VAS units minimum), number of joints (minimum of 2 worse) with active arthritis (swelling, or pain and limitation of motion), number of joints (minimum of 2 worse) with limitation of movement, erythrocyte sedimentation rate, and functional ability assessed using the disability index of the Childhood Health Assessment Questionnaire (CHAQ, 30 questions, 8 domains, 0[best]-3[worst]). Patients who withdrew or who took escape medication are classified as flared. The analysis used the Cochran-Mantel-Haenszel test with the stratification variables background use of methotrexate and oral corticosteroids applied at Week 16.
Time Frame: Week 16 through Week 40
Population: Intent-to-treat population-2: All eligible patients completing Part I of the study who were randomized into Part II of the study and received at least 1 dose of tocilizumab in Part II.
Measure: Number (95% Confidence Interval); unit: Percent of patients
Groups:
- Tocilizumab 8 or 10 mg/kg: Patients received tocilizumab 8 or 10 mg/kg intravenously every 4 weeks.
Arm/Group | Placebo | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 81 | 82
Percent of patients | 48.1 [37.0 to 59.0] | 25.6 [16.0 to 35.0]

2. Secondary Outcome: Percent of Patients Achieving Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology 30, 50, 70, and 90 (ACR30/50/70/90) Responses in Part I of the Study (Baseline to Week 16)
Description: A JIA ACR30/50/70/90 response is defined as a ≥ 30/50/70/90% response on 3 of 6 variables and no more than 1 of the remaining variables worsening > 30%. The 6 variables are physician global assessment of disease activity (20 units minimum on a 0-100 visual analog scale [VAS]), parent/patient global assessment of overall well-being (20 VAS units minimum), number of joints (minimum of 2 worse) with active arthritis (swelling, or pain and limitation of motion), number of joints (minimum of 2 worse) with limitation of movement, erythrocyte sedimentation rate, and functional ability assessed using the disability index of the Childhood Health Assessment Questionnaire (CHAQ, 30 questions, 8 domains, 0[best]-3[worst]).
Time Frame: Baseline to Week 16
Population: Intent-to-treat patient population-1: All patients who were randomized into Part I of the study and received at least 1 dose of tocilizumab.
Measure: Number; unit: Percent of patients
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 35 | 34 | 119 | 188
Percent of patients
  ACR30 response | 88.6 | 76.5 | 93.3 | 89.4
  ACR50 response | 80.0 | 70.6 | 87.4 | 83.0
  ACR70 response | 62.9 | 41.2 | 68.1 | 62.2
  ACR90 response | 31.4 | 23.5 | 25.2 | 26.1

3. Secondary Outcome: Percent Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Physician Global Assessment of Disease Activity at the End of Part I of the Study (Week 16)
Description: The patient's treating physician provides a rating of the patient's arthritis disease activity on a 0 to 100 mm horizontal scale. The extreme left end of the line represents 'arthritis inactive' (ie, symptom-free and no arthritis symptoms) and the extreme right end represents 'arthritis very active'. A higher score indicates more disease activity. A negative change score indicates improvement.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 35 | 34 | 119 | 188
Percent change | -61.48 (48.779) | -65.20 (26.170) | -72.61 (25.977) | -69.19 (31.824)

4. Secondary Outcome: Percent Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Patient/Parent Global Assessment of Overall Well-being at the End of Part I of the Study (Week 16)
Description: The patient or parent/guardian, as appropriate, provides a rating of the patient's well-being on a 0 to 100 mm horizontal scale. The extreme left end of the line represents 'very well' (ie, symptom-free and no arthritis disease activity) and the extreme right end represents 'very poor' (ie, maximum arthritis disease activity). A higher score indicates poorer well-being. A negative change score indicates improvement.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 35 | 34 | 119 | 188
Percent change | -31.65 (120.268) | -55.56 (42.092) | -53.34 (58.686) | -49.46 (72.920)

5. Secondary Outcome: Percent Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Number of Joints With Active Arthritis at the End of Part I of the Study (Week 16)
Description: Joints with active arthritis are defined as joints with swelling present or pain present and limitation of motion. The maximum number of joints with active arthritis is 71. The joint assessment is performed by an independent assessor who is not the treating physician and who is blinded to all other aspects of the patient's efficacy and safety data. A negative change score indicates improvement.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 35 | 34 | 119 | 188
Percent change | -63.36 (43.272) | -55.57 (44.876) | -72.96 (33.915) | -68.15 (38.246)

6. Secondary Outcome: Percent Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Number of Joints With Limitation of Movement at the End of Part I of the Study (Week 16)
Description: Joints with limitation of movement are defined as joints with limitation of motion. The maximum number of joints with limitation of movement is 67. The joint assessment is performed by an independent assessor who is not the treating physician and who is blinded to all other aspects of the patient's efficacy and safety data. A negative change score indicates improvement.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 35 | 34 | 119 | 188
Percent change | -61.83 (34.726) | -49.87 (48.091) | -65.96 (30.134) | -62.42 (34.955)

7. Secondary Outcome: Percent Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Erythrocyte Sedimentation Rate (ESR) at the End of Part I of the Study (Week 16)
Description: Erythrocyte sedimentation rate, an acute phase protein, was measured using a kit furnished by the study central laboratory. A negative change score indicates improvement.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 35 | 34 | 119 | 188
Percent change | -70.98 (24.530) | -21.84 (159.592) | -70.87 (33.400) | -62.54 (73.384)

8. Secondary Outcome: Percent Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Functional Ability at the End of Part I of the Study (Week 16)
Description: Functional ability is assessed with the Childhood Health Assessment Questionnaire (CHAQ-DI) disability index which consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. There are 4 possible responses to each question (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do). A domain score is the highest score in that domain. If aids and devices listed in the questionnaire or assistance from a person are required to perform a task, a domain score of 0 or 1 is increased to 2; if the domain score is 2 or 3, the domain score is not adjusted. To calculate the overall score, the patient must have a domain score in at least 6 of the 8 domains. The CHAQ-DI score is the sum of the domain scores divided by the number of domains that have a non-missing score and ranges from 0 (best) to 3 (worst). A higher score indicates less ability. A negative change score indicates improvement.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 35 | 34 | 119 | 188
Percent change | -54.48 (37.214) | -46.16 (50.961) | -49.07 (45.048) | -49.62 (44.573)

9. Secondary Outcome: Juvenile Arthritis Disease Activity Score (JADAS-27) at the End of Part I of the Study (Week 16)
Description: The JADAS-27 is derived from the following components: Physician's global assessment of disease activity on a 0-100 mm visual analog scale (VAS)/10, patient/parent's global assessment of overall well-being on a 0-100 mm VAS/10, normalized erythrocyte sedimentation rate (ESR) (if ESR is ≤ 20 then set to 0, if ≥ 120 then set to 10, and if > 20 and < 120 then apply formula [ESR-20]/10), and number of joints (maximum of 27) with active arthritis (cervical spine, left/right elbow, left/right wrist, left/right MCP1-3, left/right PIP1-5, left/right hips, left/right knee and left/right ankle). The scores for the first 3 components range from 0-10; the score for the final component ranges from 0-27. The overall JADAS-27 score ranges from 0-57. A higher score indicates more disease activity.
Time Frame: Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 35 | 34 | 119 | 188
Units on a scale | 9.08 (8.882) | 12.25 (10.277) | 7.83 (7.122) | 8.82 (8.198)

10. Secondary Outcome: Pain Visual Analogue Scale (VAS) Score at the End of Part I of the Study (Week 16)
Description: The patient or parent/guardian, as appropriate, provides a rating of the patient's pain (also called a discomfort index) on a 0 to 100 mm horizontal scale. The extreme left end of the line represents 'no pain' and the extreme right end represents 'very extreme pain'. A higher score indicates more pain.
Time Frame: Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 35 | 34 | 119 | 188
Units on a scale | 21.9 (21.66) | 24.1 (23.94) | 20.3 (21.13) | 21.2 (21.65)

11. Secondary Outcome: Percent of Patients With Inactive Disease at the End of Part I of the Study (Week 16)
Description: A patient is judged to have inactive disease if all of the following criteria are met: Number of joints with active arthritis = 0; absence of active uveitis, defined by the adverse event preferred terms 'uveitis' and 'intermediate uveitis'; normal erythrocyte sedimentation rate (< 20 mm/hour regardless of age and sex); and physician's global assessment of overall well-being visual analog scale score ≤ 10.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: Percent of patients
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 35 | 34 | 119 | 188
Percent of patients | 20.0 | 8.8 | 18.5 | 17.0

12. Secondary Outcome: Percent of Patients With an Elevated C-reactive Protein Concentration at Baseline That Had Normalized at the End of Part I of the Study (Week 16)
Description: C-reactive protein (CRP), an acute phase protein, was measured in blood samples with a high-sensitivity CRP (hs-CRP) test using laser nephelometry.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number; unit: Percent of patients
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 13 | 19 | 46 | 78
Percent of patients | 76.9 | 63.2 | 87.0 | 79.5

13. Secondary Outcome: Percent of Patients With an Elevated Erythrocyte Sedimentation Rate at Baseline That Had Normalized at the End of Part I of the Study (Week 16)
Description: Erythrocyte sedimentation rate, an acute phase protein, was measured using a kit furnished by the study central laboratory.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number; unit: Percent of patients
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 23 | 26 | 73 | 122
Percent of patients | 82.6 | 57.7 | 87.7 | 80.3

14. Secondary Outcome: Percent of Patients With an Elevated Platelet Count at Baseline That Had Normalized at the End of Part I of the Study (Week 16)
Description: Platelets were measured in blood samples taken from the patients.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number; unit: Percent of patients
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 13 | 18 | 43 | 74
Percent of patients | 84.6 | 55.6 | 86.0 | 78.4

15. Secondary Outcome: Percent of Patients With an Elevated White Blood Count at Baseline That Had Normalized at the End of Part I of the Study (Week 16)
Description: White blood cells were measured in blood samples taken from the patients.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number; unit: Percent of patients
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 3 | 3 | 2 | 8
Percent of patients | 66.7 | 66.7 | 100.0 | 75.0

16. Secondary Outcome: Percent of Patients Achieving Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology 30, 50, 70, and 90 (ACR30/50/70/90) Responses at the End of Part II of the Study (Week 40)
Description: A JIA ACR30/50/70/90 response is defined as a ≥ 30/50/70/90% response on 3 of 6 variables and no more than 1 of the remaining variables worsening > 30%. The 6 variables are physician global assessment of disease activity (20 units minimum on a 0-100 visual analog scale [VAS]), parent/patient global assessment of overall well-being (20 VAS units minimum), number of joints (minimum of 2 worse) with active arthritis (swelling, or pain and limitation of motion), number of joints (minimum of 2 worse) with limitation of movement, erythrocyte sedimentation rate, and functional ability assessed using the disability index of the Childhood Health Assessment Questionnaire (CHAQ, 30 questions, 8 domains, 0[best]-3[worst]). The analysis used the Cochran-Mantel-Haenszel test with the stratification variables background use of methotrexate and oral corticosteroids applied at Week 16.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percent of patients
Arm/Group | Placebo | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 81 | 82
Percent of patients
  ACR30 response | 54.3 [43.0 to 65.0] | 74.4 [65.0 to 84.0]
  ACR50 response | 51.9 [41.0 to 63.0] | 73.2 [64.0 to 83.0]
  ACR70 response | 42.0 [31.0 to 53.0] | 64.6 [54.0 to 75.0]
  ACR90 response | 23.5 [14.0 to 33.0] | 45.1 [34.0 to 56.0]

17. Secondary Outcome: Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Physician Global Assessment of Disease Activity at the End of Part II of the Study (Week 40)
Description: The patient's treating physician provides a rating of the patient's arthritis disease activity on a 0 to 100 mm horizontal scale. The extreme left end of the line represents 'arthritis inactive' (ie, symptom-free and no arthritis symptoms) and the extreme right end represents 'arthritis very active'. A higher score indicates more disease activity. A negative change score indicates improvement. Change from baseline was calculated using last observation carried forward imputation for missing values.
Time Frame: Baseline to Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 81 | 82
Units on a scale | -38.2 (24.77) | -45.6 (21.47)

18. Secondary Outcome: Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Patient/Parent Global Assessment of Overall Well-being at the End of Part II of the Study (Week 40)
Description: The patient or parent/guardian, as appropriate, provides a rating of the patient's well-being on a 0 to 100 mm horizontal scale. The extreme left end of the line represents 'very well' (ie, symptom-free and no arthritis disease activity) and the extreme right end represents 'very poor' (ie, maximum arthritis disease activity). A higher score indicates poorer well-being. A negative change score indicates improvement. Change from baseline was calculated using last observation carried forward imputation for missing values.
Time Frame: Baseline to Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 81 | 82
Units on a scale | -32.4 (28.57) | -31.1 (28.52)

19. Secondary Outcome: Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Number of Joints With Active Arthritis at the End of Part II of the Study (Week 40)
Description: Joints with active arthritis are defined as joints with swelling present or pain present and limitation of motion. The maximum number of joints with active arthritis is 71. The joint assessment is performed by an independent assessor who is not the treating physician and who is blinded to all other aspects of the patient's efficacy and safety data. A negative change score indicates improvement. Change from baseline was calculated using last observation carried forward imputation for missing values.
Time Frame: Baseline to Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Placebo | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 81 | 82
Joints | -11.5 (12.77) | -14.5 (11.14)

20. Secondary Outcome: Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Number of Joints With Limitation of Movement at the End of Part II of the Study (Week 40)
Description: Joints with limitation of movement are defined as joints with limitation of motion. The maximum number of joints with limitation of movement is 67. The joint assessment is performed by an independent assessor who is not the treating physician and who is blinded to all other aspects of the patient's efficacy and safety data. A negative change score indicates improvement. Change from baseline was calculated using last observation carried forward imputation for missing values.
Time Frame: Baseline to Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Placebo | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 81 | 82
Joints | -8.1 (9.90) | -10.2 (8.97)

21. Secondary Outcome: Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Erythrocyte Sedimentation Rate (ESR) at the End of Part II of the Study (Week 40)
Description: Erythrocyte sedimentation rate, an acute phase protein, was measured using a kit furnished by the study central laboratory. A negative change score indicates improvement. Change from baseline was calculated using last observation carried forward imputation for missing values.
Time Frame: Baseline to Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Placebo | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 81 | 82
mm/hour | -14.0 (28.46) | -25.2 (21.97)

22. Secondary Outcome: Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Childhood Health Assessment Questionnaire-Disability Index (CHAQ-DI) at the End of Part II of the Study (Week 40)
Description: The Childhood Health Assessment Questionnaire-Disability Index (CHAQ-DI), as a measure of functional ability, consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. There are 4 possible responses to each question (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do). A domain score is the highest score in that domain. To calculate the overall score, the patient must have a domain score in at least 6 of the 8 domains. The CHAQ-DI score is the sum of the domain scores divided by the number of domains that have a non-missing score and ranges from 0 (best) to 3 (worst). A higher score indicates less ability. A negative change score indicates improvement. Change from baseline was calculated using last observation carried forward imputation for missing values.
Time Frame: Baseline to Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 81 | 82
Units on a scale | -0.724 (0.6905) | -0.804 (0.6534)

23. Secondary Outcome: Change From Baseline in the Pain Visual Analogue Scale (VAS) Score at the End of Part II of the Study (Week 40)
Description: The patient or parent/guardian, as appropriate, provides a rating of the patient's pain (also called a discomfort index) on a 0 to 100 mm horizontal scale. The extreme left end of the line represents 'no pain' and the extreme right end represents 'very extreme pain'. A higher score indicates more pain. A negative change score indicates improvement. Change from baseline was calculated using last observation carried forward (LOCF) imputation for missing values. The analysis was adjusted for the randomization stratification factors background use of methotrexate and background use of oral corticosteroids, and the pain visual analog scale score at Baseline. The adjusted means from the fitted model are presented.
Time Frame: Baseline to Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 81 | 82
Units on a scale | -30.2 (27.12) | -31.5 (31.76)
Statistical Analysis 1: Comparison: Placebo vs Tocilizumab 8 or 10 mg/kg; Test type: Superiority or Other; ANOVA — The analysis was adjusted for the randomization stratification factors background use of methotrexate and background use of oral corticosteroids. The analysis was also adjusted for the pain visual analog scale score at Baseline; Adjusted mean - Placebo = -22.3
Statistical Analysis 2: Comparison: Placebo vs Tocilizumab 8 or 10 mg/kg; Test type: Superiority or Other; ANOVA — [p-value comment as in outcome 23, analysis 1]; Adjusted mean - Tocilizumab = -32.4
Statistical Analysis 3: Comparison: Placebo vs Tocilizumab 8 or 10 mg/kg; Test type: Superiority or Other; p = 0.0076, ANOVA — [p-value comment as in outcome 23, analysis 1]; Mean Difference (Final Values) = -10.2, 95% CI 2-sided [-17.6 to -2.7]

24. Secondary Outcome: Percent of Patients With Inactive Disease at the End of Part II of the Study (Week 40)
Description: A patient is judged to have inactive disease if all of the following criteria are met: Number of joints with active arthritis = 0; absence of active uveitis, defined by the adverse event preferred terms 'uveitis' and 'intermediate uveitis'; normal erythrocyte sedimentation rate (< 20 mm/hour regardless of age and sex); and physician's global assessment of overall well-being visual analog scale score ≤ 10.
  The statistical test is not significant due to a break in the hierarchical chain of significance testing.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percent of patients
Arm/Group | Placebo | Tocilizumab 8 or 10 mg/kg
Number analyzed (Participants) | 81 | 82
Percent of patients | 17.3 [9 to 26] | 36.6 [26 to 47]
Statistical Analysis 1: Comparison: Placebo vs Tocilizumab 8 or 10 mg/kg; The analysis used the Cochran-Mantel-Haenszel test adjusted for the randomization stratification factors background use of methotrexate and background use of oral corticosteroids; Test type: Superiority or Other; p = 1.000, Cochran-Mantel-Haenszel — 1.000 is used here as the test was considered as not significant due to the break in the hierarchical testing chain; The analysis was adjusted for the randomization stratification factors background use of methotrexate and background use of oral corticosteroids; Weighted difference = 18, 95% CI 2-sided [5 to 32]

25. Secondary Outcome: Percent of Patients Achieving Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology 30, 50, 70, and 90 (ACR30/50/70/90) Responses at Weeks 2, 52, and 104
Description: as for outcome 2
Time Frame: Week 2 to Week 104
Population: Continuous tocilizumab population: Patients randomized to tocilizumab in Part II of the study and who therefore received tocilizumab throughout the study.
Measure: Number; unit: Percent of patients
Groups:
- Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg: Patients weighing < 30 kg at baseline receiving tocilizumab 10 mg/kg whose body weight increased to ≥ 30 kg and ≥ 5 kg over baseline body weight for 3 consecutive visits had the tocilizumab dose reduced to 8 mg/kg.
- All Tocilizumab Patients: Patients received tocilizumab 8 or 10 mg/kg intravenously every 4 weeks.
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 9 | 7 | 11 | 55 | 82
Percent of patients
  Week 2 - ACR30 Response | 55.6 | 42.9 | 45.5 | 54.5 | 52.4
  Week 2 - ACR50 Response | 33.3 | 42.9 | 18.2 | 34.5 | 32.9
  Week 2 - ACR70 Response | 11.1 | 0.0 | 9.1 | 12.7 | 11.0
  Week 2 - ACR90 Response | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 52 - ACR30 Response | 100.0 | 100.0 | 100.0 | 96.4 | 97.6
  Week 52 - ACR50 Response | 100.0 | 100.0 | 90.9 | 94.5 | 95.1
  Week 52 - ACR70 Response | 100.0 | 85.7 | 72.7 | 87.3 | 86.6
  Week 52 - ACR90 Response | 88.9 | 57.1 | 54.5 | 65.5 | 65.9
  Week 104 - ACR30 Response | 100.0 | 100.0 | 90.9 | 94.5 | 95.1
  Week 104 - ACR50 Response | 100.0 | 100.0 | 90.9 | 87.3 | 90.2
  Week 104 - ACR70 Response | 88.9 | 100.0 | 90.9 | 83.6 | 86.6
  Week 104 - ACR90 Response | 88.9 | 71.4 | 72.7 | 67.3 | 70.7

26. Secondary Outcome: Percent of Patients With 4 Baseline Disease Characteristics Achieving Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology 30, 50, 70, and 90 (ACR30/50/70/90) Responses at Week 104
Description: A JIA ACR30/50/70/90 response is defined as a ≥ 30/50/70/90% response on 3 of 6 variables and no more than 1 of the remaining variables worsening > 30%. The 6 variables are physician global assessment of disease activity (20 units minimum on a 0-100 visual analog scale), parent/patient global assessment of overall well-being (20 VAS units minimum), number of joints (minimum of 2 worse) with active arthritis (swelling, or pain and limitation of motion), number of joints (minimum of 2 worse) with limitation of movement, erythrocyte sedimentation rate, and functional ability assessed using the disability index of the Childhood Health Assessment Questionnaire (CHAQ, 30 questions, 8 domains, 0[best]-3[worst]). Results are reported for the subgroups: Previous biologic treatment (yes/no), concomitant methotrexate use (yes/no), rheumatoid factor (positive/negative), concomitant oral corticosteroid use (yes/no). Last observation carried forward was applied to missing components at visits.
Time Frame: Week 104
Population: Continuous tocilizumab population: Patients randomized to tocilizumab in Part II of the study and who therefore received tocilizumab throughout the study. Patients who withdrew due to non-safety reasons are classified as non-responders. Patients who withdrew due to safety have their last available response prior to withdrawal carried forward.
Measure: Number; unit: Percent of patients
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 9 | 7 | 11 | 55 | 82
Percent of patients
  Previous Biologic Use: Yes - ACR30 (n=1,1,0,25,27) | 100.0 | 100.0 | 0.0 | 96.0 | 96.3
  Previous Biologic Use: Yes - ACR50 (n=1,1,0,25,27) | 100.0 | 100.0 | 0.0 | 80.0 | 81.5
  Previous Biologic Use: Yes - ACR70 (n=1,1,0,25,27) | 0.0 | 100.0 | 0.0 | 72.0 | 70.4
  Previous Biologic Use: Yes - ACR90 (n=1,1,0,25,27) | 0.0 | 100.0 | 0.0 | 48.0 | 48.1
  Previous Biologic Use: No - ACR30 (n=8 6,11,30,55) | 100.0 | 100.0 | 90.9 | 93.3 | 94.5
  Previous Biologic Use: No - ACR50 (n=8,6,11,30,55) | 100.0 | 100.0 | 90.9 | 93.3 | 94.5
  Previous Biologic Use: No - ACR70 (n=8,6,11,30,55) | 100.0 | 100.0 | 90.9 | 93.3 | 94.5
  Previous Biologic Use: No - ACR90 (n=8,6,11,30,55) | 100.0 | 66.7 | 72.7 | 83.3 | 81.8
  Methotrexate Use: Yes - ACR30 (n=7,7,11,42,67) | 100.0 | 100.0 | 90.9 | 95.2 | 95.5
  Methotrexate Use: Yes - ACR50 (n=7,7,11,42,67) | 100.0 | 100.0 | 90.9 | 88.1 | 91.0
  Methotrexate Use: Yes - ACR70 (n=7,7,11,42,67) | 100.0 | 100.0 | 90.9 | 83.3 | 88.1
  Methotrexate Use: Yes - ACR90 (n=7,7,11,42,67) | 100.0 | 71.4 | 72.7 | 73.8 | 76.1
  Methotrexate Use: No - ACR30 (n=2,0,0,13,15) | 100.0 | 0.0 | 0.0 | 92.3 | 93.3
  Methotrexate Use: No - ACR50 (n=2,0,0,13,15) | 100.0 | 0.0 | 0.0 | 84.6 | 86.7
  Methotrexate Use: No - ACR70 (n=2,0,0,13,15) | 50.0 | 0.0 | 0.0 | 84.6 | 80.0
  Methotrexate Use: No - ACR90 (n=2,0,0,13,15) | 50.0 | 0.0 | 0.0 | 46.2 | 46.7
  Oral Corticosteroid Use:Yes - ACR30(n=2,3,5,23,33) | 100.0 | 100.0 | 80.0 | 91.3 | 90.9
  Oral Corticosteroid Use: Yes - ACR50 (2,3,5,23,33) | 100.0 | 100.0 | 80.0 | 91.3 | 90.9
  Oral Corticosteroid Use: Yes - ACR70 (2,3,5,23,33) | 100.0 | 100.0 | 80.0 | 82.6 | 84.8
  Oral Corticosteroid Use: Yes - ACR90 (2,3,5,23,33) | 100.0 | 66.7 | 80.0 | 65.2 | 69.7
  Oral Corticosteroid Use: No - ACR30 (7,4,6,32,49) | 100.0 | 100.0 | 100.0 | 96.9 | 98.0
  Oral Corticosteroid Use: No - ACR50 (7,4,6,32,49) | 100.0 | 100.0 | 100.0 | 84.4 | 89.8
  Oral Corticosteroid Use: No - ACR70 (7,4,6,32,49) | 85.7 | 100.0 | 100.0 | 84.4 | 87.8
  Oral Corticosteroid Use: No - ACR90 (7,4,6,32,49) | 85.7 | 75.0 | 66.7 | 68.8 | 71.4
  Rheumatoid Factor: Positive - ACR30 (0,2,2,23,27) | 0.0 | 100.0 | 100.0 | 95.7 | 96.3
  Rheumatoid Factor: Positive - ACR50 (0,2,2,23,27) | 0.0 | 100.0 | 100.0 | 91.3 | 92.6
  Rheumatoid Factor: Positive - ACR70 (0,2,2,23,27) | 0.0 | 100.0 | 100.0 | 91.3 | 92.6
  Rheumatoid Factor: Positive - ACR90 (0,2,2,23,27) | 0.0 | 50.0 | 100.0 | 78.3 | 77.8
  Rheumatoid Factor: Negative - ACR30 (9,5,7,29,50) | 100.0 | 100.0 | 100.0 | 93.1 | 96.0
  Rheumatoid Factor: Negative - ACR50 (9,5,7,29,50) | 100.0 | 100.0 | 100.0 | 82.8 | 90.0
  Rheumatoid Factor: Negative - ACR70 (9,5,7,29,50) | 88.9 | 100.0 | 100.0 | 75.9 | 84.0
  Rheumatoid Factor: Negative - ACR90 (9,5,7,29,50) | 88.9 | 80.0 | 85.7 | 58.6 | 70.0

27. Secondary Outcome: Change From Baseline in the Juvenile Arthritis Disease Activity Score-71 (JADAS-71) at Week 104
Description: The JADAS-71 is composed of 4 components: Physician global assessment of disease activity on a visual analog scale (VAS) (range = 0-10, left end of the line = arthritis inactive, ie, symptom-free and no arthritis symptoms; right end = arthritis very active), patient/parent global assessment of overall well-being on a VAS (range = 0-10, left end of the line = very well, ie, symptom-free and no arthritis disease activity; right end = very poor, ie, maximum arthritis disease activity), normalized erythrocyte sedimentation rate (ESR) (range = 0-10, If ESR is ≤ 20 mm/h, set to 0. If ≥ 120 mm/h, set to 10 mm/h. If > 20 mm/h and < 120 mm/h, apply formula: [ESR - 20 mm/h]/10 mm/h), and a count of active arthritis (swelling present or pain present and limitation of motion) in 71 selected joints (range=0-71). The JADAS-71 is the sum of the 4 component scores and ranges from 0-101. A higher score indicates more arthritis disease activity. A positive change score indicates improvement.
Time Frame: Baseline to Week 104
Population: Continuous tocilizumab population: Patients randomized to tocilizumab in Part II of the study and who therefore received tocilizumab throughout the study. Only patients with non-missing data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 7 | 7 | 11 | 51 | 76
Units on a scale | -31.40 (17.471) | -24.17 (14.856) | -25.42 (13.142) | -25.70 (12.200) | -26.05 (12.941)

28. Secondary Outcome: Percent Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Physician Global Assessment of Disease Activity at Week 104
Description: The patient's treating physician provides a rating of the patient's arthritis disease activity on a 0 to 100 mm horizontal scale. The extreme left end of the line represents 'arthritis inactive' (ie, symptom-free and no arthritis symptoms) and the extreme right end represents 'arthritis very active'. A negative change score indicates improvement.
Time Frame: Baseline to Week 104
Population: Continuous tocilizumab population: Patients randomized to tocilizumab in Part II of the study and who therefore received tocilizumab throughout the study. The analysis excluded patients without a Baseline assessment or who had withdrawn.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 7 | 7 | 11 | 51 | 76
Percent change | -97.65 (2.689) | -96.01 (9.862) | -90.42 (16.306) | -87.58 (27.588) | -89.70 (23.747)

29. Secondary Outcome: Percent Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Patient/Parent Global Assessment of Overall Well-being at Week 104
Description: The patient or parent/guardian, as appropriate, provides a rating of the patient's well-being on a 0 to 100 mm horizontal scale. The extreme left end of the line represents 'very well' (ie, symptom-free and no arthritis disease activity) and the extreme right end represents 'very poor' (ie, maximum arthritis disease activity). A negative change score indicates improvement.
Time Frame: Baseline to Week 104
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 7 | 7 | 11 | 51 | 76
Percent change | -97.01 (5.323) | -38.23 (75.749) | -83.06 (25.986) | -75.81 (42.143) | -75.35 (43.779)

30. Secondary Outcome: Percent Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Number of Joints With Active Arthritis at Week 104
Description: as for outcome 5
Time Frame: Baseline to Week 104
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 7 | 7 | 11 | 52 | 77
Percent change | -98.57 (3.780) | -88.22 (24.908) | -76.43 (44.956) | -88.60 (24.043) | -87.73 (27.088)

31. Secondary Outcome: Percent Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Number of Joints With Limitation of Movement at Week 104
Description: as for outcome 6
Time Frame: Baseline to Week 104
Population: Continuous tocilizumab population: Patients randomized to tocilizumab in Part II of the study and who therefore received tocilizumab throughout the study. Each visit includes patients with a non-missing assessment at the time point. Patients who previously withdrew are excluded. Patients without a Baseline assessment are excluded.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 7 | 7 | 11 | 52 | 77
Percent change | -98.57 (3.780) | -81.81 (32.048) | -76.66 (55.781) | -79.88 (26.831) | -81.30 (31.729)

32. Secondary Outcome: Percent Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Erythrocyte Sedimentation Rate (ESR) at Week 104
Description: as for outcome 7
Time Frame: Baseline to Week 104
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 7 | 7 | 11 | 52 | 77
Percent change | -84.42 (13.141) | -89.21 (4.682) | -74.06 (31.967) | -73.85 (29.073) | -76.24 (27.263)

33. Secondary Outcome: Percent Change From Baseline in the Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Component Score Functional Ability at Week 104
Description: Functional ability is assessed with the Childhood Health Assessment Questionnaire (CHAQ-DI) disability index which consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. There are 4 possible responses to each question (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do). A domain score is the highest score in that domain. If aids and devices listed in the questionnaire or assistance from a person are required to perform a task, a domain score of 0 or 1 is increased to 2; if the domain score is 2 or 3, the domain score is not adjusted. To calculate the overall score, the patient must have a domain score in at least 6 of the 8 domains. The CHAQ-DI score is the sum of the domain scores divided by the number of domains that have a non-missing score and ranges from 0 (best) to 3 (worst). A negative change score indicates improvement.
Time Frame: Baseline to Week 104
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 7 | 7 | 11 | 52 | 77
Percent change | -96.03 (10.499) | -79.50 (18.622) | -78.58 (29.821) | -73.34 (38.745) | -76.71 (34.696)

34. Secondary Outcome: Percent of Patients With a Minimally Important Improvement in the Children's Health Assessment Questionnaire-Disability Index (CHAQ-DI) Score at Weeks 16, 40, 52, 80, and 104
Description: The CHAQ-DI consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. There are 4 possible responses to each question (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do). A domain score is the highest score in that domain. If aids and devices listed in the questionnaire or assistance from a person are required to perform a task, a domain score of 0 or 1 is increased to 2; if the domain score is 2 or 3, the domain score is not adjusted. To calculate the overall score, the patient must have a domain score in at least 6 of the 8 domains. The CHAQ-DI score is the sum of the domain scores divided by the number of domains that have a non-missing score and ranges from 0 (best) to 3 (worst). A minimally important improvement is an improvement ≥ 0.13 over Baseline. Patients who withdrew due to non-safety reasons are classified as non-responders.
Time Frame: Baseline to Week 104
Population: as for outcome 26
Measure: Number; unit: Percent of patients
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 9 | 7 | 11 | 55 | 82
Percent of patients
  Week 16 | 77.8 | 85.7 | 81.8 | 76.4 | 78.0
  Week 40 | 88.9 | 100.0 | 81.8 | 78.2 | 81.7
  Week 52 | 88.9 | 100.0 | 81.8 | 80.0 | 82.9
  Week 80 | 88.9 | 100.0 | 90.9 | 80.0 | 84.1
  Week 104 | 88.9 | 100.0 | 100.0 | 80.0 | 85.4

35. Secondary Outcome: C-reactive Protein Levels From Baseline to Week 104
Description: as for outcome 12
Time Frame: Baseline to Week 104
Population: Continuous tocilizumab population: Patients randomized to tocilizumab in Part II of the study and who therefore received tocilizumab throughout the study. Each visit includes patients with a non-missing assessment at the time point. Patients who previously withdrew are excluded.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 9 | 7 | 9 | 53 | 78
mg/L
  Week 16 (n=9, 6, 7, 53, 75) | 1.726 (2.7395) | 0.220 (0.0400) | 1.077 (1.1247) | 1.137 (3.2472) | 1.129 (2.9042)
  Week 40 (n=7, 7, 11, 51, 76) | 3.709 (9.0383) | 2.286 (5.5183) | 1.591 (2.6187) | 1.451 (5.9168) | 1.756 (5.8029)
  Week 52 (n=8, 7, 10, 52, 77) | 3.405 (8.6491) | 0.267 (0.1325) | 4.584 (10.4573) | 0.882 (2.4335) | 1.569 (5.0838)
  Week 80 (n=8, 7, 10, 51, 76) | 2.329 (5.9286) | 0.623 (0.6096) | 4.867 (13.0151) | 0.718 (1.5474) | 1.425 (5.2250)
  Week 104 (n=7, 7, 11, 50, 75) | 0.249 (0.0949) | 0.200 (0.0000) | 1.259 (2.8519) | 2.032 (6.5732) | 1.581 (5.4965)

36. Secondary Outcome: Change From Baseline in the Pain Visual Analogue Scale (VAS) Score at Weeks 2, 40, 52, and 104
Description: The patient or parent/guardian, as appropriate, provides a rating of the patient's pain (also called a discomfort index) on a 0 to 100 mm horizontal scale. The extreme left end of the line represents 'no pain' and the extreme right end represents 'very extreme pain'. A higher score indicates more pain. A negative change score indicates improvement.
Time Frame: Baseline to Week 104
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 9 | 7 | 11 | 55 | 82
Units on a scale
  Week 2 (n=9, 7, 10, 52, 78) | -11.4 (13.16) | -4.4 (13.13) | -6.1 (20.98) | -10.3 (21.44) | -9.4 (19.80)
  Week 40 (n=8, 7, 11, 52, 78) | -44.0 (12.29) | -24.7 (27.76) | -27.9 (35.85) | -33.9 (31.64) | -33.3 (30.44)
  Week 52 (n=8, 7, 1, 52, 78) | -47.8 (14.46) | -24.0 (26.59) | -29.6 (28.39) | -35.5 (29.07) | -34.9 (27.76)
  Week 104 (n=7, 7, 11, 51, 76) | -48.9 (16.71) | -30.7 (31.63) | -27.1 (39.51) | -34.5 (34.59) | -34.4 (33.72)

37. Secondary Outcome: Percent of Patients With Inactive Disease From Week 16 to Week 104
Description: A patient is judged to have inactive disease if all of the following criteria are met: Number of joints with active arthritis = 0; absence of active uveitis, defined by the adverse event preferred terms 'uveitis' and 'intermediate uveitis'; normal erythrocyte sedimentation rate (< 20 mm/hour regardless of age and sex); and physician's global assessment of overall well-being visual analog scale score ≤ 10. Patients who withdrew due to non-safety reasons are classified as non-responders.
Time Frame: Week 16 to Week 104
Population: Continuous tocilizumab population: Patients randomized to tocilizumab in Part II of the study and who therefore received tocilizumab throughout the study. Patients who withdrew due to safety have their last available response prior to withdrawal carried forward. Last observation carried forward applied to missing core components at visits.
Measure: Number; unit: Percent of patients
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 9 | 7 | 11 | 55 | 82
Percent of patients
  Week 16 | 11.1 | 42.9 | 18.2 | 20.0 | 20.7
  Week 40 | 44.4 | 42.9 | 45.5 | 38.2 | 40.2
  Week 52 | 66.7 | 57.1 | 45.5 | 50.9 | 52.4
  Week 80 | 66.7 | 57.1 | 54.5 | 56.4 | 57.3
  Week 104 | 66.7 | 71.4 | 54.5 | 63.6 | 63.4

38. Secondary Outcome: Percent of Patients in Clinical Remission From Week 40 to 104
Description: A patient was in clinical remission if they had inactive disease at all visits in the 6 months prior to and including the visit assessment day. A patient was judged to have inactive disease if all of the following criteria were met: Number of joints with active arthritis = 0; absence of active uveitis, defined by the adverse event preferred terms 'uveitis' and 'intermediate uveitis'; normal erythrocyte sedimentation rate (< 20 mm/hour regardless of age and sex); and physician's global assessment of overall well-being visual analog scale score ≤ 10. Patients who withdrew due to non-safety reasons are classified as non-responders.
Time Frame: Week 40 to Week 104
Population: as for outcome 37
Measure: Number; unit: Percent of patients
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 9 | 7 | 11 | 55 | 82
Percent of patients
  Week 40 | 0.0 | 14.3 | 0.0 | 7.3 | 6.1
  Week 52 | 22.2 | 14.3 | 18.2 | 18.2 | 18.3
  Week 80 | 55.6 | 42.9 | 36.4 | 25.5 | 31.7
  Week 104 | 55.6 | 57.1 | 27.3 | 34.5 | 37.8

39. Secondary Outcome: Percent of Patients Achieving Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology 30, 50, 70, and 90 (ACR30/50/70/90) Responses at Week 104 by Duration of Disease (< 2 Years, ≥ 2 Years)
Description: A JIA ACR30/50/70/90 response is defined as a ≥ 30/50/70/90% response on 3 of 6 variables and no more than 1 of the remaining variables worsening > 30%. The 6 variables are physician global assessment of disease activity (20 units minimum on a 0-100 visual analog scale [VAS]), parent/patient global assessment of overall well-being (20 VAS units minimum), number of joints (minimum of 2 worse) with active arthritis (swelling, or pain and limitation of motion), number of joints (minimum of 2 worse) with limitation of movement, erythrocyte sedimentation rate, and functional ability assessed using the disability index of the Childhood Health Assessment Questionnaire (CHAQ, 30 questions, 8 domains, 0[best]-3[worst]). Patients who withdrew due to non-safety reasons are classified as non-responders.
Time Frame: Baseline to Week 104
Population: as for outcome 37
Measure: Number; unit: Percent of patients
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 9 | 7 | 11 | 55 | 82
Percent of patients
  Disease Duration < 2 Years - ACR30 (n=4,1,4,17,26) | 100.0 | 100.0 | 100.0 | 88.2 | 92.3
  Disease Duration < 2 Years - ACR50 (n=4,1,4,17,26) | 100.0 | 100.0 | 100.0 | 82.4 | 88.5
  Disease Duration < 2 Years - ACR70 (n=4,1,4,17,26) | 100.0 | 100.0 | 100.0 | 82.4 | 88.5
  Disease Duration < 2 Years - ACR90 (n=4,1,4,17,26) | 100.0 | 100.0 | 100.0 | 76.5 | 84.6
  Disease Duration ≥ 2 Years - ACR30 (n=5,6,7,38,56) | 100.0 | 100.0 | 85.7 | 97.4 | 96.4
  Disease Duration ≥ 2 Years - ACR50 (n=5,6,7,38,56) | 100.0 | 100.0 | 85.7 | 89.5 | 91.1
  Disease Duration ≥ 2 Years - ACR70 (n=5,6,7,38,56) | 80.0 | 100.0 | 85.7 | 84.2 | 85.7
  Disease Duration ≥ 2 Years - ACR90 (n=5,6,7,38,56) | 80.0 | 66.7 | 57.1 | 63.2 | 64.3

40. Secondary Outcome: Oral Corticosteroid Dose at Baseline, Week 52, and Week 104
Description: Due to the different types of corticosteroid medications available, the prednisone equivalent was used in the calculation of the oral corticosteroid dose. Values are based on the average daily dose on the study day and if not available the last observation carried forward is used.
Time Frame: Baseline to Week 104
Population: All exposure safety population: All patients randomized into Part I of the study who received at least 1 infusion of tocilizumab and had at least 1 post-baseline safety assessment or event. Each visit includes patients with a non-missing assessment at the time point. Patients who previously withdrew are excluded.
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 22 | 13 | 34 | 119 | 188
mg/kg/day
  Baseline (n=22, 13, 34, 119, 188) | 0.041 (0.0704) | 0.095 (0.0836) | 0.079 (0.0802) | 0.055 (0.0708) | 0.061 (0.0743)
  Week 52 (n=17, 13, 24, 105, 159) | 0.021 (0.0474) | 0.064 (0.0599) | 0.037 (0.0591) | 0.032 (0.0490) | 0.034 (0.0518)
  Week 104 (n=16, 13, 23, 103, 155) | 0.014 (0.0418) | 0.028 (0.0497) | 0.019 (0.0412) | 0.020 (0.0558) | 0.020 (0.0518)

41. Secondary Outcome: Methotrexate Dose at Baseline, Week 52, and Week 104
Description: Values are based on the average daily dose on the study day and if not available the last observation carried forward is used.
Time Frame: Baseline to Week 104
Population: All exposure safety population: All participants randomized into Part I of the study who received at least 1 infusion of tocilizumab and had at least 1 post-baseline safety assessment or event. Each visit includes patients with a non-missing assessment at the time point. Patients who previously withdrew are excluded.
Measure: Mean (Standard Deviation); unit: mg/m^2/week
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Number analyzed (Participants) | 22 | 13 | 34 | 119 | 188
mg/m^2/week
  Baseline (n=22, 13, 34, 118, 187) | 11.304 (6.7521) | 17.562 (17.0864) | 12.146 (5.2822) | 8.768 (5.5387) | 10.292 (7.3586)
  Week 52 (n=17, 13, 24, 105, 159) | 9.247 (5.6513) | 15.568 (15.2521) | 11.216 (4.6890) | 8.326 (4.9825) | 9.453 (6.6963)
  Week 104 (n=16, 13, 23, 103, 155) | 8.342 (5.2618) | 11.858 (14.3458) | 10.050 (4.6316) | 6.855 (5.0401) | 7.902 (6.4332)

42. Secondary Outcome: Height Standard Deviation Score at Baseline, Week 52, and Week 104
Description: The height Standard Deviation Score was calculated using the following formula: (Observed height - median of the reference population)/standard deviation of the reference population. The reference population was defined as that of the same sex and age to the nearest completed year and month using the World Health Organization norms. A negative score indicates less height than the reference population.
Time Frame: Baseline to Week 104
Population: Growth population: All participants who received at least 1 dose of tocilizumab but who did not take the growth hormone somatotropin.
Measure: Mean (Standard Deviation); unit: Standard deviation score
Groups:
- Placebo to Tocilizumab: Patients received placebo to tocilizumab intravenously every 4 weeks.
Arm/Group | Placebo to Tocilizumab | Tocilizumab 8 or 10 mg/kg | All Tocilizumab Patients
Number analyzed (Participants) | 84 | 82 | 187
Standard deviation score
  Baseline | -0.57 (1.005) | -0.33 (1.290) | -0.51 (1.219)
  Week 52 | -0.51 (1.004) | -0.15 (1.216) | -0.33 (1.125)
  Week 104 | -0.34 (0.954) | -0.01 (1.150) | -0.18 (1.066)

ADVERSE EVENTS:
Time Frame: All exposure safety population: All participants randomized into Part I of the study who received at least 1 infusion of tocilizumab and had at least 1 post-baseline safety assessment or event.
Description: The patients were exposed to weight-adjusted doses for the 104 week duration of the study with the exception of those patients randomized in Part II (Weeks 16-40) to receive placebo. Adverse events (AE) are reported for all participants and by the various weight-based dose groups. AEs which occurred in the placebo group in Part II are not included.
Arm/Group | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg | All Tocilizumab Patients
Serious Adverse Events (participants affected / at risk) | 4/22 | 1/13 | 4/34 | 17/119 | 26/188
Other Adverse Events (participants affected / at risk) | 19/22 | 11/13 | 25/34 | 102/119 | 157/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg (N=22) | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg (N=13) | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg (N=34) | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg (N=119) | All Tocilizumab Patients (N=188)
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 3 | 4
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Varicella (Infections and infestations) | 1 | 0 | 1 | 0 | 2
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Cholangitis sclerosing (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Familial mediterranean fever (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 1
Uveitis (Eye disorders) | 0 | 0 | 2 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Benign intracranial hypertension (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Psychosomatic disease (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Epstein-Barr Virus Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 10 mg/kg in Patients Weighing < 30 kg (N=22) | Tocilizumab 10 mg/kg to 8 mg/kg in Patients Weighing < 30 kg (N=13) | Tocilizumab 8 mg/kg in Patients Weighing < 30 kg (N=34) | Tocilizumab 8 mg/kg in Patients Weighing ≥ 30 kg (N=119) | All Tocilizumab Patients (N=188)
Nasopharyngitis (Infections and infestations) | 7 | 1 | 5 | 32 | 45
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 4 | 17 | 23
Pharyngitis (Infections and infestations) | 4 | 1 | 3 | 18 | 26
Rhinitis (Infections and infestations) | 1 | 2 | 5 | 7 | 15
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 6 | 3 | 6 | 37 | 52
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 15 | 17
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 14 | 17
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3 | 12 | 17
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 12 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 6 | 13 | 25
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 15 | 19
Headache (Nervous system disorders) | 1 | 3 | 5 | 22 | 31
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 7 | 11
Ear infection (Infections and infestations) | 1 | 2 | 2 | 10 | 15
Gastroenteritis (Infections and infestations) | 1 | 0 | 3 | 7 | 11
Influenza (Infections and infestations) | 2 | 1 | 1 | 7 | 11
Sinusitis (Infections and infestations) | 1 | 2 | 2 | 5 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 5 | 10
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 8 | 10
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 6 | 8
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 6 | 8
Oral herpes (Infections and infestations) | 2 | 1 | 1 | 3 | 7
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0 | 6 | 7
Otitis media (Infections and infestations) | 0 | 0 | 2 | 3 | 5
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 3 | 5
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 4 | 5
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 2 | 4
Viral infection (Infections and infestations) | 0 | 1 | 0 | 3 | 4
Laryngitis (Infections and infestations) | 2 | 0 | 0 | 1 | 3
Varicella (Infections and infestations) | 1 | 2 | 0 | 0 | 3
Infection parasitic (Infections and infestations) | 0 | 1 | 1 | 0 | 2
Mumps (Infections and infestations) | 0 | 0 | 2 | 0 | 2
Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Muscle abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Skin bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 6 | 7
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 5
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 5 | 8
Rhinorrhoea (Renal and urinary disorders) | 1 | 1 | 0 | 4 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 3
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 7 | 8
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 6 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 5 | 6
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 3
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 3 | 7
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 2 | 6
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2 | 4
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 3
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 3
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 2
Conjunctivitis (Eye disorders) | 2 | 0 | 1 | 6 | 9
Iridocyclitis (Eye disorders) | 0 | 0 | 2 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2 | 6 | 8
Pyrexia (General disorders) | 0 | 1 | 2 | 4 | 7
Transaminases increased (Investigations) | 0 | 1 | 0 | 4 | 5
Hypotension (Vascular disorders) | 0 | 1 | 1 | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 2
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.